CLINICAL TRIAL: NCT02589938
Title: A Phase III Prospective Randomized Trial of Acupuncture for Treatment of Radiation-Induced Xerostomia in Patients With Head and Neck Cancer
Brief Title: Trial of Acupuncture for Radiation-Induced Xerostomia in Head and Neck Cancer
Acronym: ACUPUNCTURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IRB00038707; REBAWF 97115 (Other: NCI); NCI-2011-02073 (Registry Identifier: NCI CTRP); NCT01141231 (obsolete NCT alias)
Record Dates: First submitted 2015-08-17; First posted 2015-10-28 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Radiation-Induced Xerostomia; Head and Neck Cancer; Radiation Toxicity; Oral Complications of Chemotherapy and Head/Neck Radiation
Keywords: hypopharyngeal cancer; laryngeal cancer; lip and oral cavity cancer; nasopharyngeal cancer; oropharyngeal cancer; paranasal sinus and nasal cavity cancer; salivary gland cancer; radiation toxicity; xerostomia; long-term effects of cancer treatment; oral complications of radiation therapy
MeSH Terms: conditions — Head and Neck Neoplasms; Radiation Injuries; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Mouth Neoplasms; Nasopharyngeal Neoplasms; Oropharyngeal Neoplasms; Salivary Gland Neoplasms; Xerostomia | interventions — Oral Hygiene

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Oral Hygiene (Active Comparator): All patients will receive standard oral hygiene patient teaching information that includes instructions regarding mouth rinses, use of lip balms, use of mild fluoride toothpaste, the importance of adequate oral hydration, and other standard advice. Each participating site determines the standard oral hygiene recommendations used at their site.
  Interventions: Other: Standard Oral Hygiene
- Standard Oral Hygiene + True Acupuncture (Experimental): All patients will receive standard oral hygiene patient teaching information that includes instructions regarding mouth rinses, use of lip balms, use of mild fluoride toothpaste, the importance of adequate oral hydration, and other standard advice. Each participating site determines the standard oral hygiene recommendations used at their site.
  The True acupuncture points will be at 3 sites on each ear, a site on the chin, on each forearm, a site on each hand, a site on each leg, and one placebo needle for a total of 14 sites. All sites will be applied for 20 minutes.
  Interventions: Other: Standard Oral Hygiene + True Acupuncture
- Standard Oral Hygiene + Sham Acupuncture (Other): All patients will receive standard oral hygiene patient teaching information that includes instructions regarding mouth rinses, use of lip balms, use of mild fluoride toothpaste, the importance of adequate oral hydration, and other standard advice. Each participating site determines the standard oral hygiene recommendations used at their site.
  The Sham acupuncture points will be given according to the same schedule as the active acupuncture points, except the Sham needles will be placed below, above or between true active points.
  Interventions: Other: Standard Oral Hygiene + Sham Acupuncture

INTERVENTIONS:
Other: Standard Oral Hygiene — Oral hygiene care provided per individual institutions standard of care.
  Other Names: Oral Hygiene
  Arms: Standard Oral Hygiene
Other: Standard Oral Hygiene + True Acupuncture — Oral hygiene care provided per individual institutions standard of care. 14 true acupoint sites will be selected and applied to each participant for 20 minutes at each session. There will be 2 sessions a week for 8 weeks.
  Arms: Standard Oral Hygiene + True Acupuncture
Other: Standard Oral Hygiene + Sham Acupuncture — Oral hygiene care provided per individual institutions standard of care. 14 sham acupoint sites will be selected and applied to each participant for 20 minutes at each session. There will be 2 sessions a week for 8 weeks.
  Other Names: Placebo acupuncture needle
  Arms: Standard Oral Hygiene + Sham Acupuncture

SUMMARY:
This study is being done to find out what effects, good and/or bad, acupuncture has on participants and their xerostomia caused by radiation therapy for the treatment of the cancer.

DETAILED DESCRIPTION:
Patients who have met all eligibility criteria will be randomized to standard oral hygiene, standard oral hygiene + true acupuncture twice weekly for 4 weeks, or standard oral hygiene + sham acupuncture twice weekly for 4 weeks by a form of adaptive randomization, called minimization, because simple randomization could result in covariate imbalances .

The acupuncture points will be at three sites on each ear (Shenmen, Point Zero, Salivary Gland 2-prime), a site on the chin (CV24), a site on each forearm (Lu7), a site on each hand (LI 1-prime), a site on each leg (K6), and one placebo needle at Gb32 for a total of 14 sites. All sites will be applied for 20 minutes. For body points, standardized techniques for location will be utilized, which are based on anatomical landmarks as well as proportional measurements using the patient's own body. For example, finger breadth is based on each patient's middle finger, and the proportional unit of measure, the "cun," is defined as the distance between the two medial ends of the creases of the interphalangeal joints when the middle finger is flexed. Ear point locations will mimic standard practice and be identified by the acupuncturists.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years of age and able to give informed consent.
* Must be able to read, write and understand English.
* Must have a diagnosis of head/neck cancer.
* Must have received bilateral radiation therapy, and subsequently developed grade 2 or 3 xerostomia, according to modified Radiation Therapy Oncology Group (RTOG) scale:

  * Grade 0 - None
  * Grade 1 - Slight dryness of mouth (good response on stimulation and no significant dietary alterations necessary)
  * Grade 2 - Moderate dryness of mouth (poor response on stimulation and altered oral intake required such as frequent water, oral lubricants, or soft-moist foods)
  * Grade 3 - Complete dryness of mouth (no response on stimulation and difficult oral alimentation; IV fluids, pureed diet or tube feedings may be required)
  * Grade 4 - Fibrosis
* Must have received external beam radiation at a mean dose of at least 24 Gy to one of the parotid glands. The other gland can receive less than 24 Gy.
* Must have completed radiotherapy at least 12 months prior to entry.
* Must have anatomically intact parotid and submandibular glands. A focused (head/neck) history and exam conducted by a physician or dentist within the past year is required.
* Must be acupuncture naïve.
* Must have Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.

Exclusion Criteria:

* History of xerostomia, Sjogren's disease or other illness known to affect salivation prior to head/neck radiation.
* Suspected or known closure of salivary gland ducts on either side. (Patients addressed in inclusion criteria (i.e. those who have had one submandibular gland removed) are expected to have closure to the removed submandibular gland and will be exempt from this exclusion criteria.)
* Currently receiving or planning to use drugs, herbs, alternative medicines, or devices that could affect salivary production. Treatment known to affect salivation should be stopped at least 14 days prior to enrollment. Over the counter products used for salivary substitution are allowed, but will need to be discontinued for at least 24 hours prior to saliva and questionnaire data collection.
* Have received any investigational new drug within the past 30 days or planning to receive such during the study period.
* Active systemic infection or skin infection at or near the acupuncture sites.
* Receiving chemotherapy during study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2013-07-29 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne C Danhauer, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (36):
- United States (36):
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Queen's Medical Center, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Saint Luke's Hospital, Cedar Rapids, Iowa
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Christus Saint Vincent Regional Cancer Center, Santa Fe, New Mexico
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Meharry Medical College, Nashville, Tennessee
  - MD Anderson in The Woodlands, Conroe, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - Providence Regional Cancer System-Lacey, Lacey, Washington

IPD SHARING:
Plan to Share IPD: Yes
Wake Forest (WF) National Cancer Institute Community Oncology Research Program (NCORP) Research Base (RB) is committed to following the NIH Statement on Sharing Research Data. As of July 2018, the WF NCORP RB signed an agreement with NCI to contribute de-identified data and data dictionaries from clinical trials conducted through our RB to the NCI NCTN/NCORP data archive within 6 months of primary and non-primary publications of phase II/III and phase III trials. This will become the primary means for sharing raw data, and we will adhere to the guidelines spelled out in the National Clinical Trials Network (NCTN)/NCORP Data Archive Usage Guide. De-identified data from studies not covered by the agreement (e.g., phase II and observational studies) will be made available upon request. All data files will be de-identified. De-identification procedures will meet the HIPAA criteria as detailed in the Code of Federal Regulations, Part 45, Section 164.514.
Time Frame: 6 months after publication for a 2 year duration
Access Criteria: upon request

REFERENCES:
- [Derived] Cohen L, Danhauer SC, Garcia MK, Dressler EV, Rosenthal DI, Chambers MS, Cusimano A, Brown WM, Ochoa JM, Yang P, Chiang JS, Gordon O, Crutcher R, Kim JK, Russin MP, Lukenbill J, Porosnicu M, Yost KJ, Weaver KE, Lesser GJ. Acupuncture for Chronic Radiation-Induced Xerostomia in Head and Neck Cancer: A Multicenter Randomized Clinical Trial. JAMA Netw Open. 2024 May 1;7(5):e2410421. doi: 10.1001/jamanetworkopen.2024.10421. PMID 38739392

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was designed with first enrollment July 29,2013 under the oversight of MD Anderson (MDA) Community Clinical Oncology Program (CCOP) Research Base (RB) (NCI Division of Cancer Prevention (DCP) #MDA 04-01; MDA Protocol #2010-0547). Twenty-eight participants recruited from multiple centers. After the MDA CCOP RB was closed, the trial transferred to Wake Forest (WF) NCI Community Oncology Research Program (NCORP) RB (2UG1CA189824) where the trial continued (WF-97115) from April 2016-June 2021.
Pre-assignment Details: 258 of 281 eligible screened participants enrolled and randomized into study. Reasons for the 23 which chose not to participate: 16 no reason given 5 Too busy
  1 did not want randomization
  1 distance.
Groups:
- Standard Oral Hygiene + True Acupuncture: All patients will receive standard oral hygiene patient teaching information that includes instructions regarding mouth rinses, use of lip balms, use of mild fluoride toothpaste, the importance of adequate oral hydration, and other standard advice. Each participating site determines the standard oral hygiene recommendations used at their site.
  The True acupuncture points will be at 3 sites on each ear, a site on the chin, on each forearm, a site on each hand, a site on each leg, and one placebo needle for a total of 14 sites. All sites will be applied for 20 minutes.
  Standard Oral Hygiene + True Acupuncture: Oral hygiene care provided per individual institutions standard of care.
  14 true acupoint sites will be selected and applied to each participant for 20 minutes at each session. There will be 2 sessions a week for 8 weeks.
- Standard Oral Hygiene + Sham Acupuncture: All patients will receive standard oral hygiene patient teaching information that includes instructions regarding mouth rinses, use of lip balms, use of mild fluoride toothpaste, the importance of adequate oral hydration, and other standard advice. Each participating site determines the standard oral hygiene recommendations used at their site.
  The Sham acupuncture points will be given according to the same schedule as the active acupuncture points, except the Sham needles will be placed below, above or between true active points.
  Standard Oral Hygiene + Sham Acupuncture: Oral hygiene care provided per individual institutions standard of care.
  14 sham acupoint sites will be selected and applied to each participant for 20 minutes at each session. There will be 2 sessions a week for 8 weeks.
Period: Overall Study
Arm/Group | Standard Oral Hygiene | Standard Oral Hygiene + True Acupuncture | Standard Oral Hygiene + Sham Acupuncture
Started | 86 | 86 | 86
Completed | 62 | 73 | 69
Not Completed | 24 | 13 | 17
Not completed — Withdrawal by Subject | 11 | 5 | 6
Not completed — Lost to Follow-up | 3 | 3 | 3
Not completed — Death | 1 | 0 | 1
Not completed — Protocol Violation | 6 | 2 | 3
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Other: includes Patient found to be ineligible, distance, no benefit, lost insurance | 2 | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Oral Hygiene | Standard Oral Hygiene + True Acupuncture | Standard Oral Hygiene + Sham Acupuncture | Total
Number analyzed (Participants) | 86 | 86 | 86 | 258
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (9.2) | 65.0 (8.6) | 64.4 (9.9) | 65.0 (9.2)
Age, Customized [Count of Participants; unit: Participants]
  Age Stratification (years): <= 40 years | 0 | 0 | 2 | 2
  Age Stratification (years): 41-55 years | 16 | 14 | 13 | 43
  Age Stratification (years): 56-70 years | 46 | 50 | 47 | 143
  Age Stratification (years): > 70 years | 24 | 22 | 24 | 70
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 18 | 19 | 57
  Male | 66 | 68 | 67 | 201
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 7 | 16
  Not Hispanic or Latino | 78 | 82 | 78 | 238
  Unknown or Not Reported | 2 | 1 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 7 | 4 | 2 | 13
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 2 | 2 | 5 | 9
  White | 75 | 77 | 77 | 229
  More than one race | 0 | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 86 | 86 | 86 | 258
Insurance - Medicare [Count of Participants; unit: Participants] | 34 | 32 | 35 | 101
Insurance - Medicaid [Count of Participants; unit: Participants] | 8 | 2 | 5 | 15
Insurance - Private [Count of Participants; unit: Participants] | 47 | 56 | 51 | 154
Insurance - None [Count of Participants; unit: Participants] | 4 | 4 | 5 | 13
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.6 (6.2) | 26.0 (4.3) | 26.5 (5.7) | 26.7 (5.5)
Education [Count of Participants; unit: Participants]
  High School/GED | 20 | 18 | 17 | 55
  Some college/training | 31 | 27 | 30 | 88
  College degree (BA/BS) | 15 | 20 | 16 | 51
  Advanced degree | 10 | 11 | 13 | 34
  Unknown | 10 | 10 | 10 | 30
Job Status [Count of Participants; unit: Participants]
  Retired | 30 | 37 | 28 | 95
  Employed (FT/PT) | 31 | 29 | 26 | 86
  Disabled - unable to work | 10 | 5 | 7 | 22
  Other/Unknown | 15 | 15 | 25 | 55
Baseline values for outcomes [Mean (Standard Deviation); unit: scoring on a scale] — Self reported Xerostomia questionnaire consists of 8 items (scored on 11-point scale; 0-10). Item scores are summed and transformed linearly for final score between 0 and 80. Higher scores indicate worse xerostomia symptoms.
  The Functional Assessment of Cancer Therapy (FACT-G) Total (27 questions scored on 5-point scale; 0-4) summary score 0-108. Higher scores indicate better quality of life.
  Acupuncture Expectancy Scale (AES) is 4-item questionnaire (scored on a 5-point scale; 1-5) summary score between 4 and 20. Higher scores indicating greater expectancy. Population: Some outcome values are missing for participants at baseline
  scoring on a scale
    Xerostomia Questionnaire (XQ) Score (scale 0-80): number analyzed (Participants) | 84 | 85 | 85 | 254
    Xerostomia Questionnaire (XQ) Score (scale 0-80) | 63.2 (16.8) | 63.0 (17.1) | 62.1 (17.7) | 62.7 (17.1)
    FACT-G Total Score (scale 0-108): number analyzed (Participants) | 83 | 86 | 85 | 254
    FACT-G Total Score (scale 0-108) | 94.8 (15.9) | 98.8 (15.5) | 97.7 (15.1) | 97.1 (15.5)
    Acupuncture Expectancy Scale (AES) Score (scale 4-20): number analyzed (Participants) | 82 | 86 | 84 | 252
    Acupuncture Expectancy Scale (AES) Score (scale 4-20) | 12.7 (4.3) | 11.9 (4.1) | 11.7 (3.7) | 12.1 (4.0)

OUTCOME MEASURES:

1. Primary Outcome: Xerostomia Questionnaire Scores
Description: Self reported Xerostomia questionnaire consists of eight items (scored on an 11-point scale; 0-10), has been validated in several cohorts, and is regarded as the gold-standard measure for xerostomia.The questions are equally divided into 4 items about oral dryness while eating or chewing and 4 items about dryness while not eating or chewing. Item scores are summed and transformed linearly to produce a final summary score between 0 and 80. Higher scores represent more xerostomia. Questionnaire is completed prior to randomization and at each time point week 4, week 8, week 12, and end of study.
Time Frame: Baseline to 4, 8, 12, 26 weeks post acupuncture
Population: Intent to treat analysis. Considered and utilized all data available at each timepoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale 0-80
Arm/Group | Standard Oral Hygiene | Standard Oral Hygiene + True Acupuncture | Standard Oral Hygiene + Sham Acupuncture
Number analyzed (Participants) | 86 | 86 | 86
score on a scale 0-80
  Week 4 | 57.3 [54.0 to 60.6] | 50.6 [47.7 to 53.5] | 55.0 [52.0 to 58.0]
  Week 8 | 55.2 [51.3 to 59.1] | 48.3 [45.3 to 52.3] | 51.2 [47.6 to 54.8]
  Week 12 | 54.8 [50.9 to 58.8] | 48.9 [45.3 to 52.6] | 49.9 [46.2 to 53.7]
  Week 26 | 54.4 [50.4 to 58.4] | 49.2 [45.5 to 52.9] | 47.4 [43.6 to 51.2]
Statistical Analysis 1: Comparison: Standard Oral Hygiene vs Standard Oral Hygiene + True Acupuncture vs Standard Oral Hygiene + Sham Acupuncture; The primary endpoint was to determine whether true acupuncture (TA) was more effective than sham acupuncture (SA) or standard oral hygiene (SOH) at treating xerostomia as assessed by the xerostomia questionnaire (XQ) at Week 4. The study was powered to detect a difference of 10 points with an assumed standard deviation (SD)=16 between each pair of groups on XQ.This assumed a t-test with a two-sided significance level of 0·0133 and 84% power with 20% dropout; Test type: Superiority — Repeated measures analysis of covariance (RMANCOVA) models were constructed to assess differences in each outcome adjusting for baseline outcome value, group, time, and group by time interaction assuming an unstructured covariance. The primary objective was assessed using a linear contrast of group effect at 4 weeks; p = 0.0167, ANCOVA

2. Secondary Outcome: Functional Assessment of Cancer Therapy (FACT-G) Total
Description: The FACT-G QOL instrument discriminates between individuals with metastatic and non-metastatic disease, as well as between patients at different stages of illness. The scale has good concurrent validity, high internal consistency (0.89), and good test-re-test reliability (0.82 to 0.88). The total score is reported, which is a combination of the subscales of physical, social/family, emotional, and functional well-being, with higher scores representing better QOL. Scale range 0-108
Time Frame: Baseline, 4 , 8 , 12, and 26 weeks
Population: Intent to treat analysis. Considered and utilized all data available at each timepoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale 0-108
Arm/Group | Standard Oral Hygiene | Standard Oral Hygiene + True Acupuncture | Standard Oral Hygiene + Sham Acupuncture
Number analyzed (Participants) | 86 | 86 | 86
score on a scale 0-108
  Week 4 | 97.7 [95.8 to 99.6] | 101.6 [100.0 to 103.2] | 100.1 [98.4 to 101.8]
  Week 8 | 99.5 [97.4 to 101.6] | 101.1 [99.1 to 103.2] | 100.1 [98.2 to 102.1]
  Week 12 | 97.4 [95.5 to 99.4] | 102.1 [100.3 to 103.8] | 98.4 [96.6 to 100.2]
  Week 26 | 98.7 [96.2 to 101.1] | 100.5 [98.2 to 102.7] | 100.1 [97.8 to 102.4]

3. Secondary Outcome: The Acupuncture Expectancy Scale (AES)
Description: The 4-item AES was used to ensure there were no baseline group differences in expectations related to the benefits of acupuncture on dry mouth and to assess aspects of blinding after the first 4 weeks of acupuncture for the TA and SA groups. The AES is reliable (α=0·82) and valid by positive correlation with patient self-reported efficacy and satisfaction. The scale has been further validated among cancer patients who were acupuncture naïve. Scale from 4-20.
Time Frame: Week 4
Population: Intent to treat analysis excluding standard oral hygiene group. Considered and utilized all data available at each timepoint. AES was not collected for the standard oral hygiene arm per protocol specifications. Standard oral hygiene participants were not to receive any form of acupuncture making this outcome not applicable for these participants and therefore not collected.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale 4-20
Arm/Group | Standard Oral Hygiene + True Acupuncture | Standard Oral Hygiene + Sham Acupuncture
Number analyzed (Participants) | 86 | 86
score on a scale 4-20 | 10.8 [10.0 to 11.5] | 10.7 [9.9 to 11.5]

ADVERSE EVENTS:
Time Frame: Collected at weeks 4, 8, 12 and 24. July 29,2013 under the oversight of the MD Anderson Community Clinical Oncology Program Research Base (MDA CCOP RB) (NCI DCP #MDA 04-01; MD Anderson Protocol #2010-0547). (WF-97115) from April 2016 through June 2021.
Description: By protocol definitions, only grade 1-3 adverse events that were deemed definitely, possibly, or probably related to treatment and all grade 3-5 severe adverse events (SAEs) were to be reported.
Arm/Group | Standard Oral Hygiene | Standard Oral Hygiene + True Acupuncture | Standard Oral Hygiene + Sham Acupuncture
All-Cause Mortality (participants affected / at risk) | 1/86 | 0/86 | 1/86
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/86 | 0/86
Other Adverse Events (participants affected / at risk) | 0/86 | 3/86 | 3/86
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Oral Hygiene (N=86) | Standard Oral Hygiene + True Acupuncture (N=86) | Standard Oral Hygiene + Sham Acupuncture (N=86)
Edema face (General disorders) | 0 (0) | 0 (0) | 1 (1)
Flu like systoms (General disorders) | 0 (0) | 0 (0) | 1 (1)
Joint Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The trial was not successful at recruiting a large sample of ethnically/racially underserved participants. In addition, the majority of the patients were also men, but participation of women reflected the incidence of head and neck (HN) cancer in men and women. Most of the patients only received 4 weeks of acupuncture and no maintenance treatments were provided. Future research should examine if the effects can be enhanced with further treatments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-26): https://cdn.clinicaltrials.gov/large-docs/38/NCT02589938/Prot_SAP_001.pdf
  • Informed Consent Form (2017-08-08): https://cdn.clinicaltrials.gov/large-docs/38/NCT02589938/ICF_000.pdf